CLINICAL TRIAL: NCT00376558
Title: Imaging the Neurobiology of a Behavioral Treatment for Cocaine Dependence
Acronym: PET-CRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #5158; R01DA020855-02 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contingency Management w/ CRA (Active Comparator): Cocaine users: Contingency management w/ Community Reinforcement Approach
  Interventions: Behavioral: Community Reinforcement Approach
- Healthy Control (No Intervention): A group of healthy matched comparison subjects with no DSM-IV axis I Disorder was included; they were matched for cigarette smoking, gender, and ethnicity.

INTERVENTIONS:
Behavioral: Community Reinforcement Approach — Community Reinforcement Approach (CRA): The community reinforcement treatment program will be carried out in accordance with NIDA's therapy manual (13).During weeks 13 through 24, patients will meet once per week with their therapists. Sessions will focus on promoting continued change in the life areas addressed in the first 12 weeks of treatment or new components are added as needed.
  Arms: Contingency Management w/ CRA

SUMMARY:
The purpose of this study is to determine whether patients with the greatest loss of dopamine transmission due to cocaine dependence at pre-treatment PET and MRI scans will be those who fail to respond to substance abuse treatment. This study will also determine whether patients who do respond to treatment will experience a recovery of dopamine function. This study includes free brain imaging and behavioral intervention. Compensation provided for the brain scans.

DETAILED DESCRIPTION:
Previous studies have shown that cocaine dependence is associated with a decrease in dopamine release in response to a psychostimulant challenge. We have recently completed a study demonstrating that this loss of pre-synaptic dopamine function is associated with the choice to self-administer cocaine in the presence of an alternative reinforcer. This finding consistent with animal models of reinforcement and which show that dopamine transmission serves to modulate reward based behavior, and in this case, allows for a more adaptive response to be made in the presence of a competing reinforcer.

The previous study was performed in non-treatment seeking cocaine dependent subjects using an inpatient laboratory model to measure the choice for cocaine. Thus, the goal of the present proposal is to investigate this association in a more realistic setting where cocaine dependent out patients face the choice between using cocaine and the alternative reinforcers presented to them in a therapeutic setting. The Community Reinforcement Approach with voucher incentives is a treatment for cocaine dependence that has been shown success in a number of controlled studies. Since the basis of this therapy is to reduce the reinforcing value of cocaine by increasing the density of alternative, healthy reinforcers, we have chosen to correlate outcome from this treatment with measures of presynaptic dopamine function. We propose to scan cocaine dependent patients with [11C]raclopride and oral methylphenidate in order to measure dopamine release. Patients will be scanned before treatment and at 12 weeks into therapy. We predict that the patients with the greatest loss of dopamine transmission at the pre-treatment scan will be those who fail to respond to treatment. Furthermore, we hypothesize that the patients who do respond to treatment will experience a recovery of dopamine function, measured at the post-treatment scan.

In addition, subjects enrolled in this study will undergo functional Magnetic Resonance Imaging (fMRI) and spectroscopy studies in order to asses differences in neuronal integrity, learning, and impulse control.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 21 and 45 years old
* Fulfill DSMIV criteria for cocaine abuse or dependence
* Able to give informed consent and comply with study procedures
* Medically Healthy

Exclusion Criteria:

* Major DSM-IV Axis I disorder other than cocaine abuse or dependence. Subjects with a history of other psychostimulant abuse/dependence or compulsive gambling will be excluded.
* Current use of opiates, sedative-hypnotic, and/or cannabis more than twice a week (use less than twice a week is acceptable).
* Current use of psychotropic medication such as antipsychotics or antidepressants.
* Presence or positive history of severe medical or neurological illness (including epilepsy), or any cardiovascular disease, low hemoglobin (Hb < 14 gm/dL in males, Hb < 12 gm/dL in females), or SGOT or SGPT > 2-3 times normal. Chronic active hepatitis B or C will also be an exclusion criteria.
* Resting SBP >150, DBP > 90
* Pregnancy or lactation, lack of effective birth control during 15 days before the scans*
* Evidence /report of any heart abnormality during intake medical history, EKG or physical exam.
* Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan, as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" Shellock, PhD, Lippincott Williams and Wilkins, NY 2001.
* Lifetime exposure to radiation in the workplace, or history of participation in nuclear medicine procedures, including research protocols **
* Positive Allen Test indicating lack of collateral blood flow to hand
* History of sensitivity to methylphenidate

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, MD, Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Martinez D, Carpenter KM, Liu F, Slifstein M, Broft A, Friedman AC, Kumar D, Van Heertum R, Kleber HD, Nunes E. Imaging dopamine transmission in cocaine dependence: link between neurochemistry and response to treatment. Am J Psychiatry. 2011 Jun;168(6):634-41. doi: 10.1176/appi.ajp.2010.10050748. Epub 2011 Mar 15. PMID 21406463
- See also: Related Info — http://substanceabuse.columbia.edu/
- See also: Related Info — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Cocaine Users: Cocaine users receiving CRA
- Control Subjects: Healthy controls who undergo scans
Period: Overall Study
Arm/Group | Cocaine Users | Control Subjects
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocaine Users | Control Subjects | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (7) | 38 (6) | 37 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Binding Potential of [11C]Raclopride
Description: The relationship between Methylphenidate-induced Dopamine Release in the Striatum (Measured by Displacement of [11C]-Raclopride by Oral Methylphenidate) and Treatment Response (Measured Using Community Reinforcement Approach and Contingency Management) was studied. Dopamine Function was assessed by evaluation of endogenous Dopamine release over the course of treatment (i.e., at 3 months as compared to baseline). Endogenous Dopamine release is inversely related to the change in binding potential (delta BPND) of [11C]raclopride, in that a negative delta BPND, or increased displacement of [11C]raclopride, reflects an increase in the release of endogenous dopamine over the course of treatment.
Time Frame: baseline and 3 months
Population: Analysis for change in binding potential (binding potential difference; at baseline versus stimulant induced binding potential) was done with 24 cocaine users since one of the subjects only underwent baseline scanning. However, treatment data for all 25 cocaine users was used.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cocaine Users | Control Subjects
Number analyzed (Participants) | 24 | 25
ratio | -13.7 (8.7) | -5.8 (8.6)
Statistical Analysis 1: Comparison: Cocaine Users vs Control Subjects; Test type: Superiority or Other; p = 0.003, ANOVA

2. Secondary Outcome: Cocaine Craving, Withdrawal Symptoms, Pattern of Cocaine Use
Description: measurement of abstinence, measured as vouchers earned and clinical appointments attended using CRA
Time Frame: 2x/week for 24 weeks
Population: The number of subjects was determined from previous studies using CM/CRA
Measure: Mean (Standard Deviation); unit: dollars
Groups:
- Cocaine Abuser Undergoing CM With CRA Treatment: Participants receive voucher points for each urine sample that tested negative for benzoylecgonine. Failure to submit a scheduled sample was treated as cocaine +. Voucher points have a monetary value that can be redeemed for goods/services that are approved by the therapist. Points ($0.25) were acquired on an escalating schedule that started at 10 points for the 1st cocaine-free sample, and each subsequent cocaine-free sample increased the value by 5 points. A bonus of 40 points ($10.00) for every 3 consecutive negative sample. Abstinence was confirmed by onsite urine test (Abuscreen On-Trak system, Roche Diagnostics). Missed clinic visits and urine samples that are considered + reset the points to the initial $2.50 value and the escalation schedule resume. Submission of 5 consecutive - samples after a + urine returns the voucher points to the value prior to reset. Points earned are never lost. A maximum of $997.50 is earned for submitting negative samples at all treatment visits.
Arm/Group | Cocaine Abuser Undergoing CM With CRA Treatment
Number analyzed (Participants) | 25
dollars | 650 (0.2)
Statistical Analysis 1: Comparison: Cocaine Abuser Undergoing CM With CRA Treatment; The limbic striatum was our primary region of interest using an unpaired t test to compare BPND and deltaBPND between the treatment responders and non-responders; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; delta bpnd = -12, Standard Deviation 7

ADVERSE EVENTS:
Arm/Group | Cocaine Users | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes